CLINICAL TRIAL: NCT00833235
Title: A Natural History Study of Patients With Dry Eye
Status: Completed | Type: Observational
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Other Study IDs: MA-RES-08-001
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Lubricant Eye Drops

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tear collection
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with dry eye: No treatment is prescribed for the study. Patient dry eye progression will be followed for up to 60 months. Patients may use artificial tears to treat their dry eye symptoms.
  Interventions: Other: Artificial Tears
- Patients with no history of dry eye: No treatment is prescribed for this control group. Patients will be followed for up to 60 months. If needed, patients may use artificial tears.
  Interventions: Other: Artificial Tears

INTERVENTIONS:
Other: Artificial Tears — Artificial tears (any brand) may be used to treat dry eye symptoms.

SUMMARY:
This is a multi-center, prospective, controlled, observational study of the natural history of patients with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Males at least 55 years old or females, at least 40 years old with perimenopausal symptoms
* Baseline OSDI score of ≥ 13
* Patients with mild to moderate dry eye (dry eye disease patients only; not applicable for control group)

Exclusion Criteria:

* Use of any topical cyclosporine ophthalmic emulsion within 3 months of baseline
* History of herpes keratitis or varicella zoster keratitis
* Any history of allergic conjunctivitis
* Temporary or permanent occlusion or cauterization of the lacrimal puncta for either eye
* Any anterior segment surgery involving a limbal or corneal incision (cataract surgery), keratorefractive procedure (LASIK, LASEK, PRK) within 12 months of baseline, or expectation of such surgery within 2 years
* Patients with known systemic disease
* Any history of corneal transplant

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At least 200 dry eye patients (with at least 40% of patients with elevated biomarkers for ocular surface inflammation) will be enrolled at approximately 15-20 sites. Approximately 40-50 patients will be enrolled in the control group.
Sampling Method: Probability Sample
Enrollment: 284 (Actual)
Dates: Start 2009-02-01 (Actual); Primary Completion 2017-03-06 (Actual); Study Completion 2017-03-06 (Actual)

PRIMARY OUTCOMES:
Percentage of Patients with Progression of Dry Eye Disease | Baseline, 60 Months

SECONDARY OUTCOMES:
Change from Baseline in Ocular Surface Disease Index© (OSDI©) Score | Baseline, 60 Months
Percentage of Patients with an Increase in Blurred Vision | Baseline, 60 Months
Change from Baseline in Schirmer's Test | Baseline, 60 Months
Change from Baseline in Conjunctival Staining Score on a 6-Point Scale | Baseline, 60 Months
Change from Baseline in Corneal Staining Score on a 6-Point Scale | Baseline, 60 Months

CONTACTS AND LOCATIONS:
Overall Officials: Tes Ignacio, Study Director — Allergan
Locations (17):
- United States (17):
  - Jones Eye Institute, Little Rock, Arkansas
  - North Valley Eye Medical Group, Inc., Mission Hills, California
  - Milauskas Eye Institute, Rancho Mirage, California
  - Eye Center of Northern Colorado, Fort Collins, Colorado
  - Cape Coral Eye Center, PA, Cape Coral, Florida
  - The Eye Institute of West Florida, Largo, Florida
  - The Wilmer Eye Institute Johns Hopkins Hospital, Baltimore, Maryland
  - Minnesota Eye Consultants, P.A., Bloomington, Minnesota
  - Mulqueeny Eye Centers, Creve Coeur, Missouri
  - Mercy Eye Specilaists, Springfield, Missouri
  - Cleveland Eye Clinic, Brecksville, Ohio
  - Ophthalmic Partners Bala, Cynwyd, Pennsylvania
  - Hazleton Eye Specialists, Township, Pennsylvania
  - Vanderbilt Eye Institute, Nashville, Tennessee
  - Alkek Eye Center, Department of Ophthalmology, Houston, Texas
  - The Eye Clinic of Texas/ dba Texas Clinical Eye Research Center, League City, Texas
  - See Clearly Vision Group, McLean, Virginia

REFERENCES:
- [Derived] McDonnell PJ, Pflugfelder SC, Stern ME, Hardten DR, Conway T, Villanueva L, Hollander DA. Study design and baseline findings from the progression of ocular findings (PROOF) natural history study of dry eye. BMC Ophthalmol. 2017 Dec 28;17(1):265. doi: 10.1186/s12886-017-0646-5. PMID 29284427